CLINICAL TRIAL: NCT01382602
Title: A Double-blind, Randomized, Placebo-Controlled Study Evaluating the Safety and Effectiveness of Cook MyoSite Incorporated AMDC in Female Patients With Stress Urinary Incontinence
Brief Title: Autologous Muscle Derived Cells Female Stress Urinary Incontinence Clinical Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-019
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urinary Incontinence, Stress; Tissue Therapy (Cell Therapy); Transplantation, Autologous
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AMDC-USR (Experimental): Subjects received 1 or 2 treatments of 150 million AMDC-USR delivered via transurethral intrasphincteric injection. After completing 12 months follow-up subjects were unblinded. Subjects were followed for 2 years after initial AMDC-USR treatment.
  Interventions: Biological: AMDC-USR
- Placebo (Placebo Comparator): Subjects received 1 or 2 treatments of placebo delivered via transurethral intrasphincteric injection. After completing 12 months follow-up subjects were unblinded and could elect to receive open-label AMDC-USR treatment. Subjects that received unblinded AMDC-USR treatment were followed for 2 years after initial placebo treatment.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AMDC-USR — AMDC-USR Treatment
  Arms: AMDC-USR
Biological: Placebo — Placebo treatment
  Arms: Placebo

SUMMARY:
This is a clinical trial to study the safety and effectiveness of Autologous Muscle Derived Cells for Urinary Sphincter Repair (AMDC-USR) for the treatment of female stress urinary incontinence (SUI).

DETAILED DESCRIPTION:
Study comparing intrasphincteric injection of AMDC-USR with placebo. Subjects unblinded after 12 months visits, but followed for 2 years. Subjects randomized to placebo could elect to receive open-label AMDC-USR after completing 12 months visit.

ELIGIBILITY:
Inclusion Criteria:

* Female patient has primary symptoms of SUI, as confirmed by patient medical history and clinical symptoms, including a focused incontinence evaluation.

Exclusion Criteria:

* Patient has symptoms of pure urge incontinence as confirmed by basic evaluation of etiology from a patient medical history, including a focused incontinence history.
* Patient has symptoms of mixed urinary incontinence where urge incontinence is the predominant factor.
* Patient has had stress urinary incontinence symptoms less than 6 months prior to signing the informed consent.
* Patient has not previously attempted conservative treatment for at least 1 month prior to signing the informed consent. (Examples of conservative treatment include behavior modifications, bladder exercises, biofeedback, etc.)
* Patient has more than 2 episode of awakening to void during normal sleeping hours.
* Patient cannot be maintained on a stable dose and/or frequency of medication (including diuretics) known to affect lower urinary tract function, including but not limited to, anticholinergics, tricyclic antidepressants or alpha-adrenergic blockers, for at least 2 weeks prior to randomization or is likely to change during the course of the study.
* Patient is pregnant, lactating, or plans to become pregnant during the course of the study.
* Patient refuses to provide written informed consent.
* Patient is not at least 18 years of age.
* Patient is not available for the follow-up evaluations as required by the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-11-04 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2017-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley K. Carr, MD, FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (10):
- Canada (8):
  - Foothills Medical Center, Calgary, Alberta
  - Southern Alberta Institute of Urology, Calgary, Alberta
  - Victoria Gynecology and Continence Clinic, Victoria, British Columbia
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - Centre for Applied Urological Research Queens University, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Praxisklinik Urologie Rhein-Ruhr, Mülheim, Germany
- Worthing Hospital, Worthing, United Kingdom

REFERENCES:
- [Derived] Fontaine F, Tu LM, Carroll MS, Morin M. Agreement between simple catheter method and 3D transperineal ultrasound for assessing urethral length measurement before stress urinary incontinence treatment. Neurourol Urodyn. 2018 Nov;37(8):2875-2880. doi: 10.1002/nau.23805. Epub 2018 Sep 3. PMID 30178605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 10 sites globally; 8 sites in Canada, 1 site in Germany, and 1 site in United Kingdom.
Pre-assignment Details: 227 subjects consented to study participation and were screened for eligibility, of whom 150 subjects were enrolled (underwent biopsy procedure) and 143 subjects underwent at least 1 study treatment AMDC-USR (93 subjects) or placebo (50 subjects). Analysis population is based on 143 subjects that underwent at least 1 study treatment.
Groups:
- AMDC-USR: Subjects received 1 or 2 treatments of 150 million AMDC-USR delivered via transurethral intrasphincteric injection. After completing 12 months follow-up subjects were unblinded. Subjects were followed for 2 years after initial AMDC-USR treatment. Analysis population is based on subjects that received at least 1 treatment of AMDC-USR at the 12 months follow-up.
- Placebo: Subjects received 1 or 2 treatments of placebo delivered via transurethral intrasphincteric injection. After completing 12 months follow-up, subjects were unblinded and could elect to receive open-label AMDC-USR treatment. Subjects that received open-label AMDC-USR treatment were followed for 2 years after initial placebo treatment. Analysis population is based on subjects that received at least 1 treatment of placebo at the 12 months follow-up.
Period: Overall Study
Arm/Group | AMDC-USR | Placebo
Started | 93 | 50
Completed | 93 | 46
Not Completed | 0 | 4
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 150 subjects were enrolled and 143 subjects received at least 1 treatment of either AMDC-USR or placebo. Analysis population is based on 143 subjects that underwent at least 1 study treatment.
Groups:
- AMDC-USR: Subjects received 1 or 2 treatments of 150 million AMDC-USR delivered via transurethral intrasphincteric injection.
- Placebo: Subjects received 1 or 2 treatments of placebo delivered via transurethral intrasphincteric injection.
- Total: Total of all reporting groups
Arm/Group | AMDC-USR | Placebo | Total
Number analyzed (Participants) | 93 | 50 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 43 | 125
  >=65 years | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (11.1) | 51.7 (9.9) | 51.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 50 | 143
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 91 | 47 | 138
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 91 | 49 | 140
  United Kingdom | 1 | 0 | 1
  Germany | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response (Based on Stress IEF, or In-office Pad Weight Test, or 24-hour Pad Weight Test) at 12 Months
Description: A composite primary endpoint of responder rate was used, where a subject was considered a responder if she had ≥ 50% reduction from baseline in stress Incontinence Episode Frequency (stress IEF; reported stress leaks from 3-day diary) or ≥ 50% reduction in leakage from baseline as determined by either the in-office pad weight test or the 24-hour pad weight test.
Time Frame: 12 months
Population: Analysis population is based on subjects that received at least 1 treatment of AMDC-USR or placebo at the 12 months follow-up..
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | AMDC-USR | Placebo
Number analyzed (Participants) | 91 | 50
Percentage of subjects | 82 [73 to 90] | 90 [78 to 97]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from consent through study exit. Reporting groups are based on adverse events that occurred between initial blinded injection treatment and unblinding of subjects after 12-month follow-up.
Description: Adverse events that occurred between initial blinded injection and unblinding of subjects after 12-month follow-up were compared between AMDC-USR and Placebo groups.
Groups:
- AMDC-USR: Subjects received 1 or 2 treatments of 150 million AMDC-USR delivered via transurethral intrasphincteric injection. Analysis population is based on subjects that underwent at least 1 treatment of AMDC-USR, at the 12 month follow-up.
- Placebo: Subjects received 1 or 2 treatments of placebo delivered via transurethral intrasphincteric injection. Analysis population is based on subjects that underwent at least 1 treatment of placebo, at the 12 month follow-up.
Arm/Group | AMDC-USR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/50
Other Adverse Events (participants affected / at risk) | 32/93 | 13/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMDC-USR (N=93) | Placebo (N=50)
Urinary tract infection (Infections and infestations) | 12 | 5
Dysuria (Renal and urinary disorders) | 5 | 3
Pollakiuria (Renal and urinary disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 8 | 0
Injection site pain (General disorders) | 5 | 1

LIMITATIONS AND CAVEATS:
Planned study enrollment was 246 patients; due to limitations in study design related to the primary efficacy endpoint, enrollment was halted early at 150 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes